CLINICAL TRIAL: NCT03071016
Title: Usage of Dapagliflozin - a Sodium Glucose Co-transporter Inhibitor, in the managEment of Type-2 Diabetes Mellitus: A Real World Evidence Study in Indian Patients
Brief Title: Usage of Dapagliflozin in the Management of Type-2 Diabetes Mellitus: A Real World Evidence Study in Indian Patients
Acronym: FOREFRONT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00029
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes
Keywords: T2D,; Type 2 Diabetes,; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: None Retained — no samples retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a non-interventional, multicentre, prospective, observational study to be conducted at 50 sites in India. The study targets to enrol 2000 patients with 40 patients per site. The study will be initiated after obtaining written approval of Independent Ethics Committee (IEC) /Institutional Review Board (IRB) and written informed consent of the patient.

DETAILED DESCRIPTION:
This study is a non-interventional, multicentre, prospective, observational study to be conducted at 50 sites in India. The study targets to enrol 2000 patients with 40 patients per site. The study would enrol T2DM patients who are/were inadequately controlled (HbA1c >7%) with existing anti-diabetic medications and who have been prescribed dapagliflozin 3 months prior to study initiation. No study medication will be prescribed or administered as a part of study procedure. Patients, who have been treated as per Investigators' routine clinical practice and prescribed dapagliflozin 3 months before will be screened for enrolment in study. Dosage of dapagliflozin and other medications should be as per the routine clinical practice and prescribing information. The study will be initiated after obtaining written approval of Independent Ethics Committee (IEC) /Institutional Review Board (IRB).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with 18 years and above.
2. Patients who provide written informed consent.
3. Patients with previously diagnosed Type-2 diabetes mellitus
4. Patients with inadequately controlled diabetes (HbA1c >7%) with existing anti-diabetic medications, prior to initiation of dapagliflozin treatment.
5. Patients who are taking dapagliflozin within last 3 months.

Exclusion Criteria:

1. Patients with Type-1 diabetes mellitus
2. Patients with any medical condition which in the opinion of the investigator would interfere with safe completion of the study
3. Pregnant or lactating women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

PRIMARY OUTCOMES:
To record the mean change in HbA1C from baseline | 6 months
  form basline visit to 6 months visit

SECONDARY OUTCOMES:
To record the change in weight | 6 months
  from Baseline to 6 month visit
To record the change in blood pressure | 6 months
  from baseline to 6 month visit

CONTACTS AND LOCATIONS:
Overall Officials: Dr Vijay Viswanathan, M.D., Ph.D., FRCP, Principal Investigator — MV Hospital Chennai India
Locations (29):
- India (29):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Nellor, Andhra Pradesh
  - Research Site, Vijayawada, Andhra Pradesh
  - Research Site, Raipur, Chhattisgarh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Rajkot, Gujarat
  - Research Site, Surat, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Aurangabad, Maharashtra
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Amritsar, Punjab
  - Research Site, Bhathinda, Punjab
  - Research Site, Chandigarh, Punjab
  - Research Site, Ludhiana, Punjab
  - Research Site, Patiāla, Punjab
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Pudhucherry, Tamil Nadu
  - Research Site, Salem, Tamil Nadu
  - Research Site, Hyderabad, Telangana
  - Research Site, Kanpur, Uttar Pradesh
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Jalpāiguri, West Bengal
  - Research Site, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: D1690R00029 CSR synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4571&filename=D1690R00029_CSR_synopsis.pdf